CLINICAL TRIAL: NCT04580732
Title: Prospective, Multi-center, Randomized Trial of the MiniStim PNS for Knee Pain- "FLEX" Study
Brief Title: Clinical Trial of the MiniStim PNS for Knee Pain- "FLEX" Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MiniStim LLC (Industry)
Responsible Party: Sponsor
Organization: Uro Medical Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FLEX 31-00104
Record Dates: First submitted 2020-09-28; First posted 2020-10-08 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Chronic Knee Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active (Active Comparator): Subjects randomized to the Active group, programming parameters will be set, and therapy will be delivered for a minimum of 2-hours per day for the duration of the study.
  Interventions: Device: MiniStim PNS
- Delayed (Placebo Comparator): The delayed group will begin 2-hour stimulation/day at the 3-Month visit.
  Interventions: Device: MiniStim PNS

INTERVENTIONS:
Device: MiniStim PNS — MiniStim PNS is indicated for pain management in adults who have severe intractable chronic pain of peripheral nerve origin.

SUMMARY:
This is a prospective, multi-center, randomized, study in which 300 evaluable subjects will be randomized 1:1 to receive active or delayed therapy with Moments PNS. Subjects in the Delayed group will start with therapy at 3-month visit follow up. The primary endpoint is a >50% pain relief at 3-months as measured by the Visual Analog Scale (VAS) without increase in baseline pain medications, with additional measurements assessed at 3, 6, 9, 12, 24, and 36-months.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, multi-center study in which up to 300 evaluable subjects will receive MiniStim PNS. Target subjects will have chronic knee pain.

Subjects will be randomized into either the active or delayed group. Devices will be activated post-op in accordance to the randomization assignment. Subjects randomized to the Active group, programming parameters will be set, and therapy will be delivered for a minimum of 2-hours per day for the duration of the study. Implanted subjects will be educated on the use of the transmitter. Programming changes can be done as needed during this time period to maximize clinical response according to pre-programmed settings. Subjects randomized to the Delayed group will begin 2-hour stimulation/day at the 3-Month visit.

The primary endpoint will be at 3-Months, comparing Active vs. Delayed data from baseline data, and subjects in the Delay group will begin stimulation. At the 3-month visit, VAS will be completed and compared to baseline VAS, during this visit the safety and efficacy of the device will be assessed, and subjects in the Delayed group will be instructed to begin daily stimulation for a minimum of 2 hours a day. Subjects will be seen at 3-month intervals through the 12-Month visit for data collection and adverse event review. Subjects will continue therapy and followed for a total of 36-months with primary outcomes assessed at 3-months. Their participation in the study will end at 36-months.

ELIGIBILITY:
Inclusion Criteria:

A. Capable of giving informed consent and willing to follow all study related procedures;

B. Women and men >18 years of age;

C. Baseline VAS score of > 5;

D. History of chronic, function-limiting knee pain of at least three months;

E. Not had recent surgical procedures of the knee within the last three months;

F. ≥50% temporary relief from temporary nerve diagnostics;

G. No evidence of anatomic abnormalities that could jeopardize the placement of the device;

H. Able to operate programmer, recharger, study assessments and provide accurate responses;

I. Appropriate candidate for the implant procedure based on the opinion of investigator.

Exclusion Criteria:

A. An active implantable electronic device regardless of whether stimulation is ON or OFF;

B. Dependency on utilizing wearable or transcutaneous monitoring device (hearing aids, continuous glucose monitors, etc.);

C. Pregnant as confirmed by a urine pregnancy test or plan to become pregnant during study;

D. Subject noted no relief from temporary nerve diagnostics;

E. Inability to achieve appropriate positioning;

F. Inability to understand informed consent and protocol;

G. Conditions requiring recurring MRI evaluation or diathermy procedures;

H. Anatomical restrictions such that device placement is not possible;

I. Have a life expectancy of less than 1-year;

J. Worker's compensation claimants;

K. Based on opinion of investigator any legal concerns that would preclude his/her enrollment in the study or potentially confound results;

L. Deemed unsuitable for enrollment by investigator based on medical history or physical examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Rate of Change in Pain Relief: >50% pain relief as measured by Visual Analog Scale | 3-Months
  Improvement pain defined as a >50% pain relief as measured by VAS without increase in baseline medications. To demonstrate clinically significant improvements in the pain of subjects in the active group compared to the subjects in the delayed group.
Adverse Events | 3-months
  Device- and procedure-related Adverse Events (AE) rate at 3-months.

SECONDARY OUTCOMES:
Physical Function: Ability to do one-legged knee bends | 3, 6, 9, 12, 24, 36-months
  The ability to do one-legged knee bends (percentage increase in knee bends).
Subset Symptoms: Mental Component Score | 3, 6, 9, 12, 24, 36-months
  Change in Mental Component Score measured by SF-36 questionnaire measured on a scale of 1-5; 1 (all of the time) to 5 (none of the time).
Medication Usage | 3, 6, 9, 12, 24, 36-months
  Medication usage before and after treatment in active and delayed group subjects.
Change in Range of Motion | 3, 6, 9, 12, 24, 36-months
  Change in knee range of motion as measured with Knee Range of Motion questionnaire.
Subset Symptoms: Physical Component Score | 3, 6, 9, 12, 24, 36-months
  Change in Physical Component Score measured by SF-36 questionnaire measured on a scale of 1-5; 1 (all of the time) to 5 (none of the time).

OTHER OUTCOMES:
Change in American Knee Society Score | 3, 6, 9, 12, 24, 36-months
  Change in American Society Score before and after treatment between the treated knee and the untreated knee in active and delayed group subjects with bilateral knee pain from osteoarthritis, trauma, or surgery. The score interval is measured 0 (none) to 10 (severe).
Change in Short-Form McGill Pain Questionnaire | 3, 6, 9, 12, 24, 36-months
  Change in McGill Pain Questionnaire before and after treatment between the treated knee and the untreated knee in active and delayed group subjects with bilateral knee pain from osteoarthritis, trauma, or surgery. This questionnaire is measured on a scale of 0 (none) to 10 (worst possible).
Change in Western Ontario and McMaster University Arthritis Index | 3, 6, 9, 12, 24, 36-months
  Change in Western Ontario and McMaster University Arthritis Index before and after treatment between the treated knee and the untreated knee in active and delayed group subjects with bilateral knee pain from osteoarthritis, trauma, or surgery. The Western Ontario and McMaster University Arthritis Index scale is measured on a scale of 1 (none) to 5 (extreme).
Change in Global Perceived Effect Scales | 3, 6, 9, 12, 24, 36-months
  Change in Global Perceived Effect Scales (GPES) before and after treatment between the treated knee and the untreated knee in active and delayed group subjects with bilateral knee pain from osteoarthritis, trauma, or surgery. The Global Perceived Effect Scales range is measured from 1 (much worse) to 7 (much better).
Change in Quality of Life | 3, 6, 9, 12, 24, 36-months
  Change in Quality of Life (QoL) captured utilizing on the EQ-5D-5L survey, the form captures quality of life activities such as Mobility, Self-Care, Usual Activities, Pain/Discomfort, and rating their health for the day from 0 to 100. The EQ-5D-5L survey is measured from having no problems, slight problems, moderate problems, severe problems, or unable to perform quality of life activities.
Change in Douleur Neuropathique 4 Questionnaire | 3, 6, 9, 12, 24, 36-months
  Change in Douleur Neuropathique 4 questionnaire to estimate the degree of neuropathic pain before and after treatment in active and delayed group subjects, minimum score of 1 and maximum score of 10.
Work Status | 3, 6, 9, 12, 24, 36-months
  Work history and status will be evaluated based on a subject's self-reported questionnaire(s) completed at screening/baseline and all follow up visits.
Operating time, skin to skin and irradiation time | 3, 6, 9, 12, 24, 36-months
  Operating time, skin-to-skin time, and irradiation time for implant surgery will be collected and tallied in each treatment group.
Pain Location maps | 3, 6, 9, 12, 24, 36-months
  Pain location maps will be developed for each subject at baseline and follow-up to document and evaluate area of pain throughout the study.
Safety Assessment: Adverse Events | 6, 9, 12, 24, 36 months
  Device- and procedure-related Adverse Events (AE) rate throughout the study

CONTACTS AND LOCATIONS:
Locations (1):
- Seva Medical, Lewisville, Texas, United States